CLINICAL TRIAL: NCT03491631
Title: A Phase I Study to Characterize the Tolerance, Safety, Pharmacokinetics/Pharmacodynamics and Effect of PD-1 Inhibitor SHR-1210 in Combination With IDO Inhibitor SHR9146 and With/Without Apatinib in Patients With Advanced Solid Tumors (PIANO)
Brief Title: Phase I Study of SHR9146 + SHR-1210 +/- Apatinib in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SHR9146-I-101
Record Dates: First submitted 2018-04-01; First posted 2018-04-09 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Tumor, Solid; Cancer, Metastatic; Neoplasm Malignant
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 drugs combination group (Experimental)
  Interventions: Drug: SHR9146+SHR-1210
- 3 drugs combination group (Experimental)
  Interventions: Drug: SHR9146+SHR-1210+Apatinib

INTERVENTIONS:
Drug: SHR9146+SHR-1210 — SHR9146: Initial dose of 100mg BID with escalation planned to 600mg BID; SHR-1210: 200mg Q2W
  Arms: 2 drugs combination group
Drug: SHR9146+SHR-1210+Apatinib — SHR9146: Initial dose of 100mg BID with escalation planned to 600mg BID; SHR-1210: 200mg Q2W Apatinib:250mg QD
  Arms: 3 drugs combination group

SUMMARY:
This phase I trial is designed to efficiently identify the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) for the combination therapy regimen of the IDO1 inhibitor SHR9146 when administered in combination with immune checkpoint PD-1 inhibitor SHR-1210 plus VEGFR inhibitor Apatinib or not in subjects with advanced/metastatic solid tumors. All subjects will receive the same standard SHR-1210 plus Apatinib (only three drugs group)regimen, while SHR9146 in doses increasing from 100 mg twice daily to, potentially, 600 mg twice daily. Once the recommended regimen has been identified, subjects with the selected tumor type will be enrolled into expansion cohorts based upon prior safety and tolerability data.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically or cytologically confirmed advanced or metastatic solid tumors that have failed prior standard therapy (including subject refusal or intolerance).
2. At least one measurable parameter according to RECIST 1.1.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
4. Life expectancy of at least 12 weeks.
5. Subjects must have normal organ and marrow function as defined below:

   1. Absolute neutrophil count > 1,500/mcL
   2. Platelets > 100,000/mcL
   3. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN); for subjects with liver metastases, Total bilirubin≤ 2 x ULN,
   4. AST/ALT (SGOT/SGPT) ≤ 2.5 times institutional normal limits; for subjects with liver metastases, ALT and AST ≤ 5 × ULN
   5. Creatinine ≤ 1.5 times the ULN
6. Subjects with known brain metastases will only be eligible after their tumors have been treated with definitive resection and/or radiotherapy and they are neurologically stable for at least two months apart and at least 1 month off steroids.
7. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Known history of hypersensitivity to any components of SHR9146 and SHR-1210 formulation, or other antibody formulation.
2. Prior exposure to any T cell co-stimulatory therapy or immune checkpoint inhibitors, including but not limited to other anti-CTLA-4, anti-PD-1, anti-PD-L1 and anti-PD-L2 antibodies.
3. Prior systemic chemotherapy, radiotherapy, immunotherapy, hormone therapy, surgery or target therapy within 4 weeks (Or 5 half-life of the drug, calculate the longer ) before the study drug administration, or any unresolved AEs > Common Terminology Criteria for Adverse Events (CTCAE) Grade 1.
4. Patients with any active autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatitis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Asthma that requires intermittent use of bronchodilators or other medical intervention should also be excluded.
5. Active brain metastasis or meningeal metastasis.
6. Clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, or coronary artery bypass surgery, Congestive heart failure (New York heart association (NYHA) class > 2), ventricular arrhythmia which need medical intervention.
7. Any other medical, psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results.
8. Severe or uncontrolled systemic disease such as clinically significant hypertension(systolic pressure >/= 140 mm Hg and/or diastolic pressure >/= 90 mm Hg). (group 2)
9. Previous digestive tract bleeding history within 3 months or evident gastrointestinal bleeding tendency, such as: esophageal varices, local active ulcerative lesions, gastric ulcer and duodenal ulcer, the ulcerous colitis, gastrointestinal diseases such as portal hypertension or resection of tumor with bleeding risk, etc. (group 2)
10. Previous Arterial/venous thrombosis events within 3 months. (group 2)
11. Proteinuria ≥ (++) or 24 hours total urine protein > 1.0 g. (group 2)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
DLT | Baseline through 27/28 days
MTD | Baseline through 27/28 days

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, Prof., Principal Investigator — Jilin Provincial Tumor Hospital
Locations (1):
- Jilin Province Cancer Hospital, Changchun, Jilin, China